CLINICAL TRIAL: NCT05549089
Title: The Validity of Customized Orthodontic Bracket Set up (Randomized Clinical Trial)
Brief Title: The Validity of Customized Orthodontic Bracket Set up
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ammar Alubaydi (Other)
Responsible Party: Sponsor-Investigator, Ammar Alubaydi, clinical and lab investigator (orthodontist, PhD student), University of Baghdad
Organization: University of Baghdad (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 624422
Record Dates: First submitted 2022-09-13; First posted 2022-09-22 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Orthodontic Appliance Complication
Keywords: digital and manual orthodontic setup; customized orthodontic bracket; indirect bonding tray

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CAD/CAM Insignia™ brackets (Experimental): The result from this group (10 patients) considered as a gold standard for other two groups through assessing the treatment outcomes using American Board of Orthodontics (ABO) scoring.
  Interventions: Device: Insignia™ twin brackets
- Software-driven indirect bonding tray (Experimental): The first comparison group (10 patients): digital setup, virtual bracket placement and creation of 3D printing indirect bounding tray by using Maestro® 3D Ortho Studio software.
  Interventions: Device: Maestro® 3D Ortho Studio software (Discovery, Dentaurum®, Ispringen, Germany)
- Manual-driven indirect bonding tray (Experimental): the second comparison group (10 patients): digital setup by using Maestro® 3D Ortho Studio software, but the bracket positioning done manually by using Ray Set® device. in this group using double-layer vacuum-formed thermoplastic indirect bonding tray.
  Interventions: Device: Ray set® device (Discovery, Dentaurum®, Ispringen, Germany)

INTERVENTIONS:
Device: Insignia™ twin brackets — it is metal orthodontic twin brackets with customized base and individual arch-wires for each patient
  Arms: CAD/CAM Insignia™ brackets
Device: Maestro® 3D Ortho Studio software (Discovery, Dentaurum®, Ispringen, Germany) — it is conventional metal orthodontic twin brackets will be customizing the bracket base with adhesive composite, individual arch-wires for each patient and 3D printing indirect bonding tray
  Arms: Software-driven indirect bonding tray
Device: Ray set® device (Discovery, Dentaurum®, Ispringen, Germany) — it is conventional metal orthodontic twin brackets will be customizing the bracket base with adhesive composite, individual arch-wires for each patient and double-layer vacuum-formed thermoplastic indirect bonding tray
  Arms: Manual-driven indirect bonding tray

SUMMARY:
CAD/CAM systems have assisted orthodontists in planning and positioning brackets to minimize errors and improve the excellence of treatment. This study aimed to validate measurements obtained from manual and digital systems, as well as evaluate the effectiveness, and periodontal changes that occurred after the treatment. Materials and Methods: This study is a prospective randomized controlled trial, in which clinical evaluation of virtual setup (digital and manual) techniques versus CAD/CAM brackets (Ormco© Insignia™ .022" twin brackets) in terms of expression of bracket prescription and treatment outcome. The sample consisted of 30 young adults with Angle Class I malocclusion. Cone beam computer tomography (CBCT) were obtained before and after the treatment to assess the parallelism between the dental roots and periodontal conditions. Digital impression by three dimensional (3D) intraoral scans (IOS) will be obtained for all participants. The 3D models are converted to stereolithography (STL) for all groups. The sample will be dividing randomly into three groups; the first one treated with CAD/CAM brackets (Ormco© Insignia™ .022" twin brackets), while the other two groups were treated by customization of bracket base of the conventional pre-adjusted twin bracket with orthodontic adhesive material, this will be done through planning and creating the virtual setup by using Maestro® 3D Ortho Studio software. The Indirect bonding devices for the second group will manufacturing from 3D printed models while third group from the manual double-layer vacuum-formed thermoplastic trays. All patients will treat with fixed orthodontic twin brackets appliances. The 3D models of the Virtual setup are comparing with the treated occlusion. The linear and angular measurements are performing by the Geomagic® software and using the 3Shape's Ortho-Analyzer TM software in all groups to assess the American Board of Orthodontics grading system scores. Random errors are assessing by Intra-class Correlation Coefficient (ICC) and method errors. Descriptive statistical analysis, Shapiro-Wilk test to detect the normality of variable distribution and the Chi-square test evaluated whether the ABO scores measurements are within the limits of agreement of each criterion. ABO scores between both groups are analyze by using Wilcoxon test. The Bland-Altman analysis evaluated if differences are within the limits of agreement.

DETAILED DESCRIPTION:
Introduction Treatment efficiency has become an increasingly important goal of orthodontic treatment, yet basic questions about the efficiency of bracket system remain. In contemporary preadjusted edgewise orthodontic appliance, the greatest challenge in the success of orthodontic therapy depends undoubtedly on the perfection in bracket design, prescription, and its positioning in addition to the orthodontist's skill and training. However, due to uneven and dissimilar tooth surface anatomy, the need for an accurate method of bracket positioning with pre-determined torque and angulation incorporated in the brackets according to the patients' need is of key importance.

Therefore, it is valuable to know, dose digital bracket setting offers better outcomes? Previously, indirect bracket positioning technique was done using plaster dental cast where kesling setting (teeth alignment) made using the clinical crown. However, recently digital technique was used to assess teeth setting and bracket positioning acknowledging root positioning using typodonts.

Null hypothesis:

There is no difference between the CAD/CAM brackets setting technique (Ormco© Insignia™ .022" twin brackets) and virtual (digital and manual) bracket setting technique regarding to treatment efficiency and root positioning.

Aim and Objectives: The aim of the present study is to compare the efficacy of the virtual digital / manual setup technique compared to indirect bonded CAD/CAM brackets (Insignia™ twin brackets) in terms of expression of bracket prescription and treatment outcome using American Board of Orthodontics (ABO) scoring.

Primary Objectives: The bracket positional accuracy between manual setup-model indirect bonding and digital-driven indirect bonding methods.

Secondary Objectives: Determine the incidence of bracket debonding rate. Methodology Study design: This study is a prospective randomized controlled trial, in which clinical evaluation of virtual setup (digital and manual) techniques versus CAD/CAM brackets (Ormco© Insignia™ .022" twin brackets) in terms of expression of bracket prescription and treatment outcome.

Sample size: All patients will be recruited from the multicenter with one operator. Prior to initiating recruitment, a convenient sample size will be recruited. Initially the effect size in the sense of Cohen's for the material effect will be determined based on a previous study to be about 0.69. It was determined that the current study would reach 0.80% power with a total sample size of 54 dental arches, given that the type I error is 0.05.

Methods: Patients fulfill the selection criteria are recruited at their case presentation appointment, and consent form will be obtained. All patients informed to take CBCT before and after orthodontic treatment. The 30 consecutive patients (10 in each group) will be divided randomly into the virtually digital (Maestro® 3D Ortho Studio software) setup, manual (Ray set® device) setup and the CAD/CAM digitally (insignia®) customized group.

In this study will be use orthodontic adhesive to customize twin brackets base (Discovery, Dentaurum, Ispringen, Germany) for both manual and digital (Maestro® 3D Ortho Studio software) groups and CAD/CAM brackets (Insignia™ twin brackets) for 3rd group. On the day of recruitment, a baseline (T0) three-dimensional (3D) intraoral scan (IOS) will be done for the CAD/CAM all groups.

Manual indirect bonding setups and digital setups will be processed, as will be described in the laboratory setting section, for all teeth apart of the second molars according to previous study and verified using an objective grading system (OGS) of American Board of Orthodontics (ABO), which is currently the gold standard for evaluating plaster casts of completed orthodontic cases. In the ABO-OGS, there are eight criteria, seven of which are occlusal (tooth alignment, vertical positioning of marginal ridges, overjet, occlusal relationship, buccolingual inclination of posterior teeth, occlusal contacts, and interproximal contacts) that assess on plaster models to evaluate a patient's final occlusion. The remaining last criteria is root angulation measured on CBCT. After setups approval, indirect bonding trays or jigs will be constructed and divided randomly to the patients. After completion of bonding, an intraoral scanner will be taken to compare the bracket positioning.

Each patient received the same treatment protocol i.e., wire gauges and visiting intervals, type of ligation and finishing procedure. At the time of bracket bonding the patients will undergo an intraoral scan for the 1st and 2nd group (T1). At the working phase a 0.019*0.25 stainless steel wire will be inserted for 8 weeks, and the patients will undergo an intraoral scan (T2) and sent for CBCT.

No stopping guidelines will be specified, since subjects were receiving the same treatment materials as they would receive as part of standard care of clinical treatment. Bracket types will not blind in this study, since clear visual difference exists between the two bonding techniques, however, after bonding the treatment will be double blind for person who work on the superimposing software and statistician.

After obtaining all intraoral scans, Best-fit superimpositions will be performed depending on palatal rugae, which have been shown to be stable landmarks for the upper arch while in the lower arch, second molars (which were not engaged with Arch-wires) are used as stable landmarks.

1. ST GROUP: Manually bracket base customization:

   In the first group of this study, the stone dental cast will undergo to step wise procedure in bracket positioning and fabricating an indirect bonding tray for labial orthodontics using the Ray set device®:
2. ND GROUP: Software-driven indirect bonding Set-Up: The dental arch will undergo to a digital scanning procedure by intraoral scanner. After scanning, the digital models are sending to software-driven bracket placement.
3. RD GROUP: Insignia TM system:

The Approver Guide provides a suggested process for reviewing your Insignia cases. Having a systematic approach should save time, improve consistency, and help you manage cases more efficiently.

Scanning final Bonded Bracket positions: The final bonded bracket positions will be scanned with the intraoral scanner for the 1st and 2nd groups. This scan acquired the exact locations of the brackets bonded to the patient's teeth. This acquired image of the final bracket position will be superimposed with the initial virtual model in order to compare the bonding accuracy of the evaluated methods.

Superimposition of the digitized models: The STL files of the brackets placed using the Maestro® 3D Ortho Studio software will be exported along with the STL files of the scans of the brackets bonded intraorally.

The superimposition process consisted of defining, manually, three points for each model to superimpose (tripod), along with a precise automatic system that allowed the alignment and superimposition of the selected three points of reference. Lastly, the software will identify differences in bracket placement between the two different indirect bonding systems.

Methods of measurement before and after indirect bonding transfer:

The Geomagic control X software was used to measure the mesio-distal translation difference (in mm), the bucco-lingual translation difference (mm) and the occluso-gingival translation difference (mm) between the virtually planned brackets (STL files from the Maestro® 3D Ortho Studio software) and the brackets bonded intraorally (STL files from the intraoral scans). Each virtually planned bracket will be aligned with the origin of the three-dimensional coordinate system at the center-point of an imaginary rectangle constructed on the profile of the bracket's four wings and with the z-axis passing through the long axis of the bracket and the x-axis passing through the center of the bracket's slot.

The same method is used for the intraorally scanned brackets, where center-point Zero will be maintained as the point of reference. On the two superimposed brackets, the mesio-distal translation difference is measured by calculating the distance between the z-axis of the virtually planned bracket with a point passing perpendicular to the z-axis of the bracket scanned intraorally. In the same way, the occluso-gingival translation difference will be measured by calculating the distance between the x-axis of the virtually planned bracket with a point passing perpendicular to the x-axis of the bracket scanned intraorally.

To measure the bucco-lingual difference, the virtually planned bracket will be aligned with center-point Zero of an imaginary rectangle constructed on the profile of the two bracket wings, with the y-axis perpendicular to the long axis of the bracket, and the x-axis passing through the center-point of the rectangle, parallel to the slot base. On the basis of the two superimposed brackets, the bucco-lingual difference is measured by calculating the difference between the x-axis of the virtually planned bracket and an orthogonal point passing through the x-axis of the bracket scanned intraorally.

Evaluation of mesiodistal tip and labiolingual torque outcomes of manually and virtual-driven orthodontic appliances:

1. A pre-treatment digital model (pre-model) =pre-treatment IOS for clinical crown with pre-treatment CBCT scan and a post-treatment digital model (post-model) = post-treatment IOS for clinical crown with post treatment CBCT scan of a patient will be retrieved from the database.

   The virtual model resulting from the pre-CBCT/pre-model superimposition represents the "expected root position" (ERP) setup; it is defined as a prediction of the three-dimensional position of the roots after the orthodontic treatment
2. The virtual model resulting from superimposing and combining the post-CBCT, and the post-model represents the "true root position" (TRP) setup, as the post-CBCT depicts the three-dimensional position of the roots.
3. Each tooth isolated from the pre-treatment digital model (pre-model) is individually exported using the STL file format, in order to be superimposed independently onto the post-treatment digital model (post-model) by using software ''best fit alignment'' to overlay the teeth. Color code representing differences between the setup models.
4. In order to assess the accuracy of the iterative closest point superimposition, color maps are generated to visualize the distribution and the extent of the changes occurred between ERP and TRP.
5. The ERP and TRP STL files are then imported into software to calculate angular distances between ERP and TRP. Reference landmarks in linear measurements will be identified on the root apexes of incisors and canines; the buccal root is evaluated for premolars, the palatal root for maxillary molars, and the distal root for lower molars. The center of the angle between the root apexes of the ERP and the TRP will be identified on the crown of the post-model; it is located on the mesial incisal edge of incisors, on the tip of the vestibular cusp of canines and premolars, on the tip of the mesial cusp of maxillary molars, and on the tip of the distal cusp of mandibular molars.

Statistical Analysis:

Descriptive statistics will be presented, and data distribution will be assessed. Accordingly parametric and nonparametric statistics will be used. A P-value of <0.05 will be set to define the statistical level. Intra-observer error will calculate using an Intra-class Correlation Coefficient (ICC).

ELIGIBILITY:
Inclusion Criteria:

* Class 1 malocclusion.
* Non-extraction treatment plan.
* Initial Little Index between 5-10 mm.
* Presence of all permanent teeth.

Exclusion Criteria:

* Any systemic diseases such as diabetes, hypertension.
* Sound or clicking in temporomandibular joint or craniofacial syndromes.
* Periodontal disease or pockets greater than 4mm.
* Incisor mandibular plane angle (IMPA) ≥ 100 degrees; or any anterior tooth completely blocked from the arch form

Ages: 15 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2022-06-03 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-09-12 (Actual)

PRIMARY OUTCOMES:
American Board of Orthodontics (ABO) scoring | 18 months
  scoring system consist of 8 items:
  1. Alignment, 2. Marginal ridge height, 3. Buccolingual inclination, 4. Overjet, 5. Occlusal contacts, 6. Occlusal relationships, 7. Interproximal contacts (1-7) Component: scores < 0.5 = 0. 0.5 to 1 mm =1. > 1 mm = 2. 8. Root angulation: Root parallelism = 0. Roots are not parallel = 1. Contacting adjacent tooth = 2. High scores on individual segments, or combinations of individual segments, may cause a case to become Incomplete.
  SO:
  the minimum value = 0 the maximum value = 16 the high score means = worse outcome the low score means = better outcome

SECONDARY OUTCOMES:
linear and angular measurement of the bracket position | 4 months
  The bracket positional accuracy between manual setup-model indirect bonding and digital-driven indirect bonding methods. This done by superimposition of actual bracket position on virtual bracket position by using Geomagic® Control X™

CONTACTS AND LOCATIONS:
Overall Officials: Dheaa H Al-Groosh, phd, Principal Investigator — collage of dentistry- Baghdad university; Ammar S Alubaydi, MSc, Study Chair — collage of dentistry- Baghdad university
Locations (1):
- collage of dentistry-Baghdad university, Baghdad, Iraq

REFERENCES:
- [Derived] Al-Ubaydi AS, Al-Groosh D. Do the Various Indirect Bonding Techniques Provide the Same Accuracy for Orthodontic Bracket Placement? (Randomized Clinical Trial). Int J Dent. 2024 Jan 22;2024:5455197. doi: 10.1155/2024/5455197. eCollection 2024. PMID 38288393